CLINICAL TRIAL: NCT07151885
Title: The Diagnostic Value of Subharmonic Imaging Technology Combined With Liver Stiffness and Platelet Count for High-risk Esophageal and Gastric Varices in Patients With Liver Cirrhosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-MS-306
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices
Keywords: Liver Cirrhosis; Esophageal and Gastric Varices; Subharmonic Aided Pressure Estimation
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices

STUDY DESIGN:
Intervention Model Description: This study proposes for the first time a multimodal model integrating SHAPE, LSM and PLT, aiming to overcome the shortcomings of traditional tools, improve the prediction accuracy of high-risk EGV, and provide a new path for optimizing non-invasive screening strategies.
Masking Description: The SHAPE operator and the analyst, the LSM operator, and the gastroscopy operator blinded each other (unaware of each other's results and clinical data), and the SHAPE images were independently analyzed by two ultrasound physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHAPE (Experimental): Use an ultrasound probe to scan the liver to locate the portal vein and hepatic vein. In the angiography mode, the portal vein and hepatic vein of the same depth were selected for measurement respectively. Ultrasound contrast agent was injected through the elbow vein to observe the changes of sub-harmonic signals in the portal vein and hepatic vein. Collect the sub-harmonic signal data of the portal vein and hepatic vein, and calculate the difference between the two, that is, the SHAPE gradient.
  Interventions: Diagnostic Test: SHAPE

INTERVENTIONS:
Diagnostic Test: SHAPE — Use an ultrasound probe to scan the liver to locate the portal vein and hepatic vein. In the angiography mode, the portal vein and hepatic vein of the same depth were selected for measurement respectively. Ultrasound contrast agent was injected through the elbow vein to observe the changes of sub-harmonic signals in the portal vein and hepatic vein. Collect the sub-harmonic signal data of the portal vein and hepatic vein, and calculate the difference between the two, that is, the SHAPE gradient.

SUMMARY:
To evaluate the diagnostic value of the combined model of subharmonic-assisted pressure estimation (SHAPE), liver stiffness (LSM), and platelet count (PLT) for high-risk esophageal and gastric varices (HRV)

ELIGIBILITY:
Inclusion Criteria:

* ① Be at least 18 years old② Clinically diagnosed as liver cirrhosis (based on medical history, physical signs, laboratory tests, imaging or liver biopsy)③ Underwent a gastroscopy④ The informed consent form has been signed

Exclusion Criteria:

* ① Previous EV bleeding or having received TIPS/ endoscopic treatment.② History of concurrent liver cancer, portal vein thrombosis, and splenectomy.③ Having used drugs that affect platelet count, liver function or coagulation function in the body within one week, and having a recent history of blood product infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
HV-PV (dB) | Within two weeks of admission
  The difference in the average harmonic signal between the hepatic vein and the portal vein
Measurement of liver stiffness（kPa） | Within two weeks of admission
  The patient lies on their back, with their right hand placed behind their head. The right upper limb is fully abducted to expose the intercostal Spaces in the right lobe of the liver. The area usually enclosed by the horizontal line of the xiphoid process, the midline of the right axilla and the lower edge of the rib is taken as the testing area. The probe is vertically and closely attached to the skin, and the measurement position is selected in the intercostal space.
blood platelet count（×10⁹／L） | Within two weeks of admission
  The peripheral blood of the patient was tested by a conventional blood analyzer to obtain the platelet count.
sensitivity and specificity | The one-year period from enrollment to the end of the group
  The sensitivity measures the ability of the model to correctly identify patients with HRV (i.e., the true positive rate), and the specificity measures the ability of the model to correctly exclude patients without HRV (i.e., the true negative rate).
Positive predictive value (PPV) and negative predictive value (NPV) | The one-year period from enrollment to the end of the group
  PPV represents the probability that patients identified as high-risk by the model actually have HRV, while NPV represents the probability that patients identified as low-risk by the model do not actually have HRV
AUC | The one-year period from enrollment to the end of the group
  Comprehensively reflect the overall discriminative ability of the model under different thresholds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Wang H, Wen B, Chang X, Wu Q, Wen W, Zhou F, Guo Y, Ji Y, Gu Y, Lai Q, He Q, Li J, Chen J, Hou J. Baveno VI criteria and spleen stiffness measurement rule out high-risk varices in virally suppressed HBV-related cirrhosis. J Hepatol. 2021 Mar;74(3):584-592. doi: 10.1016/j.jhep.2020.09.034. Epub 2020 Oct 8. PMID 33039403
- [Background] Ding NS, Nguyen T, Iser DM, Hong T, Flanagan E, Wong A, Luiz L, Tan JY, Fulforth J, Holmes J, Ryan M, Bell SJ, Desmond PV, Roberts SK, Lubel J, Kemp W, Thompson AJ. Liver stiffness plus platelet count can be used to exclude high-risk oesophageal varices. Liver Int. 2016 Feb;36(2):240-5. doi: 10.1111/liv.12916. Epub 2015 Sep 6. PMID 26212020
- [Background] Vorobioff JD, Groszmann RJ. Prevention of portal hypertension: from variceal development to clinical decompensation. Hepatology. 2015 Jan;61(1):375-81. doi: 10.1002/hep.27249. Epub 2014 Sep 26. PMID 24913395
- [Background] Stefanescu H, Marasco G, Cales P, Fraquelli M, Rosselli M, Ganne-Carrie N, de Ledinghen V, Ravaioli F, Colecchia A, Rusu C, Andreone P, Mazzella G, Festi D. A novel spleen-dedicated stiffness measurement by FibroScan(R) improves the screening of high-risk oesophageal varices. Liver Int. 2020 Jan;40(1):175-185. doi: 10.1111/liv.14228. Epub 2019 Sep 11. PMID 31444849
- [Background] Yu S, Chen W, Jiang Z. Platelet count/spleen volume ratio has a good predictive value for esophageal varices in patients with hepatitis B liver cirrhosis. PLoS One. 2021 Dec 2;16(12):e0260774. doi: 10.1371/journal.pone.0260774. eCollection 2021. PMID 34855845
- [Background] Diaz-Soto MP, Garcia-Tsao G. Management of varices and variceal hemorrhage in liver cirrhosis: a recent update. Therap Adv Gastroenterol. 2022 Jun 20;15:17562848221101712. doi: 10.1177/17562848221101712. eCollection 2022. PMID 35757384
- [Background] Liang H, Si H, Liu M, Yuan L, Ma R, Zhang G, Yang J, Mo Z, Zhao Q. Non-Invasive Prediction Models for Esophageal Varices and Red Signs in Patients With Hepatitis B Virus-Related Liver Cirrhosis. Front Mol Biosci. 2022 Jul 12;9:930762. doi: 10.3389/fmolb.2022.930762. eCollection 2022. PMID 35911970
- See also: Related Info — https://linkinghub.elsevier.com/retrieve/pii/S0168827821022996
- See also: Liang H, Si H, Liu M, et al. Non-invasive prediction models for esophageal varices and red signs in patients with hepatitis B virus-related liver Cirrhosis[J]. Frontiers in Molecular Biosciences, 2022, 9: 930762. — https://www.frontiersin.org/articles/10.3389/fmolb.2022.930762/full
- See also: Yu S, Chen W, Jiang Z. Platelet count/spleen volume ratio has a good predictive value for esophageal varices in patients with hepatitis B liver Cirrhosis[J]. PLOS One, 2021, 16(12): e0260774. — https://dx.plos.org/10.1371/journal.pone.0260774
- See also: Vorobioff J D, Groszmann R J. Prevention of portal hypertension: From variceal development to clinical Decompensation[J]. Hepatology, 2015, 61(1): 375～381. — https://journals.lww.com/01515467-201501000-00043
- See also: ] De Franchis R, Bosch J, Garcia-Tsao G, et al. Baveno VII - renewing consensus in portal Hypertension[J]. Journal of Hepatology, 2022, 76(4): 959～974. — https://linkinghub.elsevier.com/retrieve/pii/S0168827821022996